CLINICAL TRIAL: NCT01952171
Title: The International Genetic Basis of Congenital Heart Disease Study
Brief Title: The Genetic Basis of Congenital Heart Disease in Africa
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: University of Lagos, Nigeria (Other); Uganda Heart Institute (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913207; 13-HG-N207
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-07-03

CONDITIONS: Congenital Heart Disease; Heart Disease
Keywords: Genomics; Birth Defects; Congenital Heart Disease; Natural History
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital Heart Disease: Congenital Heart Disease

SUMMARY:
Recent advances in genomic techniques are making possible a new wave of genetic discovery in congenital heart disease (CHD). Existing data suggests that CHD occur in Sub-Saharan Africa at frequencies similar to the rest of the world. In this application, we propose to utilize the unique advantages of Sub-Saharan Africa - a combination of the most genetically diverse populations in the world and of diminished environmental background effects (i.e. low prevalence of smoking, alcohol abuse, obesity in comparison to western countries) - to better understand the genetic basis for congenital heart disease. We will couple next generation genomic techniques with more traditional gene discovery methods to investigate CHD in two African countries: Uganda and Nigeria. The inclusion of syndromic and non-syndromic CHD observed in these populations as well as careful phenotyping (including echocardiography) will greatly enhance our potential to provide insight into the genetic architecture of CHD in African populations. To accomplish this, we plan to enroll families, in whom members have congenital heart malformations consistent with an error of early human development in our research protocol. Patients will be enrolled at the Uganda Heart Institute in Kampala, Uganda, and at the Department of Pediatrics, College of Medicine, University of Lagos, Nigeria, with the potential to include other African sites. High throughput genomic studies will be done at the NIH....

DETAILED DESCRIPTION:
Recent advances in genomic techniques are making possible a new wave of genetic discovery in congenital heart disease (CHD). Existing data suggests that CHD occur in Sub-Saharan Africa at frequencies similar to the rest of the world. In this application, we propose to utilize the unique advantages of Sub-Saharan Africa - a combination of the most genetically diverse populations in the world and of diminished environmental background effects (i.e. low prevalence of smoking, alcohol abuse, obesity in comparison to western countries) - to better understand the genetic basis for congenital heart disease. We will couple next generation genomic techniques with more traditional gene discovery methods to investigate CHD in two African countries: Uganda and Nigeria. The inclusion of syndromic and non-syndromic CHD observed in these populations as well as careful phenotyping (including echocardiography) will greatly enhance our potential to provide insight into the genetic architecture of CHD in African populations. To accomplish this, we plan to enroll families, in whom members have congenital heart malformations consistent with an error of early human development in our research protocol. Patients will be enrolled at the Uganda Heart Institute in Kampala, Uganda, and at the Department of Pediatrics, College of Medicine, University of Lagos, Nigeria, with the potential to include other African sites. High throughput genomic studies will be done at the NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study will include affected individuals and their affected/or unaffected family members. Family members will include parents and siblings. The goal will to be obtaining a minimum of a trio (affected and both parents) to increase probability of finding gene mutations. Clinical criteria for inclusion is defined as presence of a congenital cardiac malformation related to errors in early human development. The diagnosis of congenital heart disease (presence of a congenital cardiac malformation thought to be related to errors in early human development) will be made by a cardiologist on our team based on echocardiogram (performed by C.S., A.B. or E.E.), physical examination, medical history, and review of medical record.

EXCLUSION CRITERIA:

Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.

Ages: 1 Month to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include affected individuals and their affected/or unaffected family members. Family members will include parents and siblings. The goal will to be obtaining a minimum of a trio (affected and both parents) to increase probability of finding gene mutations. Clinical criteria for inclusion is defined as presence of a congenital cardiac malformation related to errors in early human development. The diagnosis of congenital heart disease (presence of a congenital cardiac malformation thought to be related to errors in early human development) will be made by a cardiologist on our team based on echocardiogram, physical examination, medical history, and review of medical record.
Sampling Method: Non-Probability Sample
Enrollment: 1233 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Genetic Diagnosis | One patient visit only
  The primary outcome is a genetic diagnosis for congenital heart disease. There are no treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Adebowale A Adeyemo, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States
- College of Medicine, University of Lagos, Lagos, Nigeria
- Chiang Mai University, Chiang Mai, Thailand

REFERENCES:
- [Derived] Ekure EN, Adeyemo A, Liu H, Sokunbi O, Kalu N, Martinez AF, Owosela B, Tekendo-Ngongang C, Addissie YA, Olusegun-Joseph A, Ikebudu D, Berger SI, Muenke M, Han Z, Kruszka P. Exome Sequencing and Congenital Heart Disease in Sub-Saharan Africa. Circ Genom Precis Med. 2021 Feb;14(1):e003108. doi: 10.1161/CIRCGEN.120.003108. Epub 2021 Jan 15. PMID 33448881